CLINICAL TRIAL: NCT05893147
Title: BALANCE+: A Platform Trial for Gram Negative Bloodstream Infections
Brief Title: BALANCE+ Vanguard Phase
Acronym: BALANCE+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4369
Record Dates: First submitted 2023-05-18; First posted 2023-06-07 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Gram-negative Bacteremia

STUDY DESIGN:
Intervention Model Description: 72 in the overall platform AND at least 12 in each domain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- De-escalation VS No De-escalation (Active Comparator)
  Interventions: Other: De-escalation VS No De-escalation
- Oral beta-lactams VS Oral Non-beta-lactams (Active Comparator)
  Interventions: Other: Oral beta-lactams VS non beta-lactams
- Central vascular catheter retention VS Central vascular catheter replacement (Active Comparator)
  Interventions: Other: Central vascular catheter retention VS Central vascular catheter replacement
- Cephalosporin VS Carbapenem for low risk AmpC organisms (Active Comparator)
  Interventions: Other: Cephalosporin VS Carbapenem for low risk AmpC organisms
- Routine follow-up blood culture VS No routine follow-up blood culture (Active Comparator)
  Interventions: Other: Routine follow-up blood culture VS No routine follow-up blood culture

INTERVENTIONS:
Other: De-escalation VS No De-escalation — No de-escalation group: continue to receive the same antibiotic that was started initially (as long as it is confirmed to be effective based on the blood culture sensitivity result)
  De-escalation group: switched to narrower spectrum antibiotic.
  Arms: De-escalation VS No De-escalation
Other: Oral beta-lactams VS non beta-lactams — Beta-lactam antibiotic: This can be ciprofloxacin, moxifloxacin, levofloxacin or trimethoprim-sulfamethoxazole.
  Non beta-lactam antibiotic: This can be, but not limited to, amoxicillin, amoxicillin-clavulanate, cephalexin, cefadroxil, or cefixime.
  Arms: Oral beta-lactams VS Oral Non-beta-lactams
Other: Central vascular catheter retention VS Central vascular catheter replacement — Central vascular catheter replacement: the catheter will be changed by the treating team as soon as possible and within a maximum of 72 hours from blood culture finalization
  Central vascular catheter retention: the catheter will not be changed and will be retained until it is no longer needed.
  Arms: Central vascular catheter retention VS Central vascular catheter replacement
Other: Cephalosporin VS Carbapenem for low risk AmpC organisms — Cephalosporin (ceftriaxone) at standard doses
  Carbapenem (like Meropenem, Ertapenem etc) at standard doses
  Arms: Cephalosporin VS Carbapenem for low risk AmpC organisms
Other: Routine follow-up blood culture VS No routine follow-up blood culture — Routine follow-up blood culture: routine repeat blood collection 4 days from the index blood collection with positive bacteria.
  No follow-up blood culture: no routine repeat blood collection 4 days from the index blood collection with positive bacteria
  Arms: Routine follow-up blood culture VS No routine follow-up blood culture

SUMMARY:
The goal of the BALANCE+ clinical trial is to transform random care to randomized care for patients with Gram negative bloodstream infections to inform best treatment approaches and optimize outcomes.

BALANCE+, a perpetual platform trial, will efficiently answer multiple questions that are important for hospitalized patients with Gram negative bloodstream infections.

DETAILED DESCRIPTION:
Bloodstream infections (BSIs) are common and lethal, ranking among the top 7 causes of death, with 600,000 cases and 90,000 deaths per year in North America, and 1.2 Million cases and 150,000 deaths per year in Europe. Despite being a leading cause of death worldwide, bloodstream infections remain understudied. Treatment approaches are complicated by rising rates of antimicrobial resistance and declining new drug development.

BALANCE+ provides a platform upon which to answer multiple pressing cross-cutting questions for patients with Gram negative bloodstream infections, including the concept of de-escalating antibiotic spectrum, optimal transition to oral antibiotics, and the role for routine follow up blood culture testing. The trial will also include a syndrome-specific question of whether to remove or retain a central vascular catheter, and a pathogen-specific question of whether cephalosporins are sufficient for patients with low-risk AmpC organisms. As each question is answered, optimal therapies will be adopted into usual care, and new questions will be introduced into the platform of the trial. The evidence generated by BALANCE+ will improve cure for this vulnerable patient population.

ELIGIBILITY:
PLATFORM INCLUSION CRITERIA

1. admitted to a participating hospital
2. positive blood culture with Gram negative (GN) bacterium

PLATFORM EXCLUSION CRITERIA

1. patient's goals of care are for palliation with no active treatment
2. moribund patient, not expected to survive > 72 hours

DOMAIN SPECIFIC INCLUSION AND EXCLUSION CRITERIA

(A) DE-ESCALATION VS. NO DE-ESCALATION DOMAIN

Inclusion Criteria

1. included in BALANCE+ platform

Exclusion Criteria

1. receiving an empiric antibiotic regimen at the time of blood culture finalization to which the GN pathogen(s) are not sensitive
2. carbapenem-resistance (so that patients will not need to remain on reserve-use agents)
3. no de-escalation option due to any or all of

   i. resistance ii. allergies iii. medical contraindications iv. drug-interaction risk v. other relevant reason
4. patients with a suspected or proven polymicrobial source of infection

(B) BETA-LACTAM VS. NON-BETA-LACTAM ORAL/ENTERAL TREATMENT DOMAIN

Inclusion Criteria

1. included in BALANCE+ platform
2. initially treated with intravenous antibiotics, but clinical team transitioning patient to oral/enteral antibiotic within 7 days of starting treatment

Exclusion Criteria

1. enrolled in an arm of another BALANCE+ platform domain which limits the use of oral/enteral therapy

   - no-de-escalation arm
2. no non-beta-lactam options due to any or all of

   i. resistance ii. allergies iii. medical contraindications iv. drug-interaction risk v. other relevant reason
3. no beta-lactam options due to any or all of

   i. resistance ii. allergies iii. medical contraindications iv. drug-drug interaction risk v. other relevant reason

(C) CENTRAL VASCULAR CATHETER REPLACEMENT DOMAIN

Inclusion Criteria

1. included in BALANCE+ platform
2. has an indwelling central vascular catheter that was already in place within the 48-hour period before the onset of bloodstream infection (i.e. is not a new catheter placed within 48 hours of the onset of infection)

Exclusion Criteria

1. patient has no ongoing need for a central vascular catheter
2. patient has definite indication for central vascular catheter removal

   1. ongoing septic shock with definite/probable line source
   2. concomitant S. aureus bacteremia
   3. concomitant candidemia
   4. local suppurative signs (severe redness, warmth, pain, swelling or fluctuance/collection) necessitating catheter removal, or other clinical evidence of infected line (e.g. imaging/echocardiographic findings)
   5. definite alternative source of GN BSI

(D) LOW-RISK AmpC DOMAIN

Inclusion Criteria

1. included in BALANCE+ platform
2. positive blood culture with GN bacterium, of the following species

   1. Serratia spp.
   2. Morganella spp.
   3. Providencia spp.
   4. Proteus spp. other than P.mirabilis
   5. organism is sensitive to ceftriaxone

Exclusion Criteria

1. severe allergy to beta-lactams (eg, type 4 hypersensitivity reaction or DRESS)
2. baseline phenotypic resistance to ceftriaxone

(E) FOLLOW UP BLOOD CULTURE DOMAIN

Inclusion Criteria

1. included in BALANCE+ platform

Exclusion Criteria

1. patient already discharged home prior to day 4
2. definite indication for repeat blood culture testing

   1. concomitant Staph. aureus bacteremia
   2. concomitant Candidemia
   3. clinical suspicion for infective endocarditis (e.g., presence of prosthetic valve, implantable cardiac device)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2023-08-26 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Recruitment rate (co-primary outcomes of BALANCE+ vanguard phase) | 1 year
  Recruitment rate will be measured as the number of patients randomized to each study domain, overall, and by individual participating site. Investigators will target a minimum overall recruitment rate of 1 patient/site/month in the de-escalation domain, beta-lactam versus non-beta-lactam stepdown domain, and FUBC domain; and 0.25 patients/site/month in the line replacement domain.
Protocol adherence (co-primary outcomes of BALANCE+ vanguard phase) | 1 year
  Protocol adherence will be calculated differently depending on the domain, but in each case will require adherence to the specific intervention arm and complete follow-up for the primary outcome. Investigators will target ≥90% adherence in each arm of each domain.
De-escalation versus no de-escalation domain | 90 days
  * Patient-centered, ordinal Desirability of Outcome Ranking (DOOR) outcome: (dead at 90 days) < (alive at 90 days with reinfection and readmission) < (alive at 90 days with reinfection or readmission) < (alive at 90 days with neither reinfection nor readmission)
  * Tie-breaker within ordinal levels: new antimicrobial resistance (AMR) colonization or infection from routine cultures
Oral beta-lactam versus non beta-lactam domain | 90 days
  * Ordinal DOOR outcome: (dead at 90 days) < (alive at 90 days with reinfection and readmission) < (alive at 90 days with reinfection or readmission) < (alive at 90 days with neither reinfection nor readmission)
  * Tie-breaker within ordinal levels: new AMR colonization or infection from routine cultures
Central vascular catheter retention versus replacement domain | 90 days
  * Ordinal DOOR outcome: (dead at 90 days) < (alive at 90 days with reinfection and readmission) < (alive at 90 days with reinfection or readmission) < (alive at 90 days with neither reinfection nor readmission)
  * No tie-breaker
Low-risk AmpC domain | 90 days
  * Ordinal DOOR outcome: (dead at 90 days) < (alive at 90 days with reinfection and readmission) < (alive at 90 days with reinfection or readmission) < (alive at 90 days with neither reinfection nor readmission)
  * Tie-breaker within ordinal levels: new AMR colonization or infection from routine cultures
Follow-up blood culture domain | 90 days
  * Ordinal DOOR outcome: (dead at 90 days) < (alive at 90 days with reinfection and readmission) < (alive at 90 days with reinfection or readmission) < (alive at 90 days with neither reinfection nor readmission)
  * No tie-breaker

SECONDARY OUTCOMES:
90-day mortality | 90 days
90-day reinfection | 90 days
90-day all cause readmission | 90 days
90-day AMR colonization/infection | 90 days
90-day Clostridioides difficile infection (CDI) | 90 days
30-day mortality | 30 days
60-day mortality | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Nick Daneman, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Rob Fowler, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (10):
- Canada (10):
  - Foothills Hospital, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Eastern Regional Health Authority, St. John's, Newfoundland and Labrador
  - The Ottawa Hospital, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - North York General Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daneman N, Johnstone J, Lee TC, MacFadden DR, McDonald EG, Morpeth SC, Ong SWX, Paterson DL, Pinto RL, Rishu A, Rogers BA, Yahav D, Coburn B, Daley P, Das P, Fiest K, Findlater A, Fralick M, George M, Kandel C, Malavade A, Powis J, Somayaji R, Fowler R; BALANCE+ Investigators, and the Association of Medical Microbiology and Infectious Disease Canada Clinical Research Network and the Canadian Critical Care Trials Group. Assessing the feasibility of a platform trial for Gram negative bloodstream infections: results from the vanguard phase of BALANCE. BMJ Open. 2025 Dec 5;15(12):e101588. doi: 10.1136/bmjopen-2025-101588. PMID 41360461